CLINICAL TRIAL: NCT02450279
Title: Scintigraphic Comparison of Lung Deposition With Two Nebulizers During Invasive Mechanical Ventilation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Never started
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AeroVent-02
Record Dates: First submitted 2015-05-18; First posted 2015-05-21 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2016-12

CONDITIONS: Post-operative Neurosurgery
Keywords: Aerosol delivery; Invasive mechanical ventilation; Jet Nebulizer; Vibrating-Mesh nebulizer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Nebulization with a vibrating-mesh nebulizer (Active Comparator): Nebulization performed with a vibrating-mesh nebulizer
  Interventions: Drug: technetium-99m - Diethylenetriaminepentaacetic acid; Device: Vibrating-mesh nebulizer; Other: Planar scintigraphy; Other: Preoperative spirometry
- Nebulization with a jet nebulizer (Active Comparator): Nebulization performed with a jet nebulizer
  Interventions: Drug: technetium-99m - Diethylenetriaminepentaacetic acid; Device: Jet Nebulizer; Other: Planar scintigraphy; Other: Preoperative spirometry

INTERVENTIONS:
Drug: technetium-99m - Diethylenetriaminepentaacetic acid
Device: Vibrating-mesh nebulizer
  Arms: Nebulization with a vibrating-mesh nebulizer
Device: Jet Nebulizer
  Arms: Nebulization with a jet nebulizer
Other: Planar scintigraphy
Other: Preoperative spirometry

SUMMARY:
Many devices are available for nebulising drug solution during invasive mechanical ventilation. Vibrating-mesh nebulizers ensure the highest lung deposition output. A recent international survey on aerosol therapy during mechanical ventilation (Ehrmann et al. 2013) reported that jet nebulizers remained the mostly used.

The aim of this study is to compare lung deposition of a radiolabeled administered with both nebulizers during invasive mechanical ventilation by planar scintigraphy.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation
* Healthy lungs

Exclusion Criteria:

* Discontinued procedure due to adverse events.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
Pulmonary deposition | Immediately after nebulization by imaging assessment, an expected average of 30 minutes

SECONDARY OUTCOMES:
Penetration index | Immediately after nebulization by imaging assessment, an expected average of 30 minutes
Mechanical ventilation settings | During nebulisation time, an expected average of 15 minutes
Lung function | Preoperative assessment, the day before inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-François Laterre, Study Chair — Head of Intensive Care Unit, Cliniques Universitaires Saint-Luc
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium